CLINICAL TRIAL: NCT01642524
Title: The Toronto Prehospital Hypertonic Resuscitation-Head Injury and Multi Organ Dysfunction Trial
Brief Title: The Toronto Prehospital Hypertonic Resuscitation Head Injury and Multi Organ Dysfunction Trial (TOPHR HIT)
Acronym: TOPHR HIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Defence Research and Development Canada (Industry)
Responsible Party: Principal Investigator, Dr. Laurie Morrison, Clinician Scientist, Unity Health Toronto
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TOPHR HIT
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Traumatic Brain Injury
Keywords: resuscitation
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypertonic saline mixed Dextran (Experimental): hypertonic saline mixed Dextran
  Interventions: Biological: hypertonic saline mixed Dextran
- Placebo controlled (Placebo Comparator): Saline solution
  Interventions: Biological: Saline solution

INTERVENTIONS:
Biological: hypertonic saline mixed Dextran — single dose administered intravenously
  Arms: hypertonic saline mixed Dextran
Biological: Saline solution — placebo - saline solution
  Arms: Placebo controlled

SUMMARY:
The TOPHR HIT trial is a clinical trial of patients experiencing blunt trauma who present with an injury to their head which makes them unconscios. The study compares two different fluids given to the patient in the out of hospital setting by a paramedic. The two fluids are salt water (standard treatment) versus a higher concentration of salt water mixed with a sugar (study fluid). The patients have an equal chance of receiving either fluid and the paramedic and the patient and the treating trauma surgeon do not know which fluid was provided in the out of hospital setting.

DETAILED DESCRIPTION:
Study Objective

The primary objective of this study is to report feasibility in accordance with the methodology described by Lancaster and Dodds, specifically addressing:

1. baseline survival rates for the treatment and control group to aid in the design of a definitive multicentre trial.
2. randomization compliance rate.
3. ease of protocol implementation in the out-of-hospital setting.
4. adverse rate of Hypertonic Saline Dextran (HSD) infusion.

The secondary objectives include measuring the effect of HSD in modulating the immuno-inflammatory response to severe head injury and its effect on modulating the release of neuro-biomarkers into serum; evaluating the role of serum neuro-biomarkers in predicting patient outcome and clinical response to HSD intervention; evaluating effects of HSD on brain atrophy post-injury and neurocognitive and neuropsychological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16
* Initial assessment of Glasgow Coma Score (GCS) 8 or less
* Blunt traumatic mechanism of injury

Exclusion Criteria:

* Known pregnancy
* Penetrating primary injury
* VSA prior to randomization; previous intravenous therapy ≥ 50 ml
* Time interval between arrival at scene and intravenous access exceeds four hours
* Amputation of above wrist or ankle
* Any burn (thermal, chemical, electrical, radiation)
* Suspected hypothermia
* Asphyxia (strangulation, hanging, choking, suffocation, drowning) and fall from height ≤ 1m or ≤ 5 stairs.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2004-04; Primary Completion 2006-01 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
30 day survival | 30 days after discharge

SECONDARY OUTCOMES:
Survival | 48 hrs after admission
  •Survival: 48 hours after admission; Hospital discharge
Functional neurological outcomes at 4 months | 4 Months
Neuropsychological testing at 4 months | 4 months
Neuropsychological testing at 1 year | 1 year
Physiologic parameters indicative of organ dysfunction | 4 months
Structural parameters indicative of brain injury or dysfunction at 4 months | 4 months
Serum inflammatory markers measured on arrival, 12, 24, 48 hours later | 12, 24, 48 hours later